CLINICAL TRIAL: NCT01280552
Title: A Randomized, Double-blind, Controlled Phase IIb Study of the Safety and Efficacy of ICT-107 in Newly Diagnosed Patients With Glioblastoma Multiforme (GBM) Following Resection and Chemoradiation
Brief Title: A Study of ICT-107 Immunotherapy in Glioblastoma Multiforme (GBM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Precision Life Sciences Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ICT-107-201
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICT-107 (Experimental): Autologous dendritic cells pulsed with immunogenic peptides from tumor antigens
  Interventions: Biological: ICT-107
- Control (Placebo Comparator): Autologous dendritic cells that have not been pulsed with antigens
  Interventions: Biological: Placebo DC

INTERVENTIONS:
Biological: ICT-107 — Autologous dendritic cells pulsed with immunogenic antigens
  Arms: ICT-107
Biological: Placebo DC — Autologous dendritic cells (DC) that have not been pulsed with antigens
  Arms: Control

SUMMARY:
This is a phase 2, multicenter study to determine the safety and efficacy of ICT-107 in treating a type of brain tumor called Glioblastoma Multiforme (GBM). ICT-107 is an immunotherapy in which the patient's immune response will be stimulated to kill the tumor cells. Patients must be newly diagnosed with GBM and not yet received chemoradiation. Some of the patient's white blood cells (WBC) will be removed and cultured in a laboratory with purified antigens, similar to those on GBM cells. The patient's own WBC/DC that have been exposed to the tumor antigens will then be given back to the patient as a vaccine over several months. The goal is for the ICT-107 vaccine to stimulate the patient's immune response to kill the remaining GBM tumor cells after surgery and chemotherapy.

DETAILED DESCRIPTION:
The proposed phase 2 study is a randomized, double blind, controlled study of the safety and efficacy of ICT-107 in newly diagnosed patients with glioblastoma multiforme (GBM) following resection and chemoradiation. The phase 1 clinical trial demonstrated safety and promising efficacy in a small, open-label study. The purpose of this study is to provide information from a larger, controlled clinical trial. Patients must be newly diagnosed with GBM and not yet received chemoradiation. Patients will have had tumor resection, magnetic resonance imaging (MRI) and tumor assessment prior to enrollment into the study. Post surgical treatment consists of 6 weeks of chemotherapy (TMZ) and radiation followed by a washout period. After Screening and informed consent, patients will undergo apheresis at the study site for collection of peripheral blood mononuclear cells (PBMCs). Apheresis product will be sent to a central site where monocytes will be purified and cultured into dendritic cells (DC). DC will be pulsed with synthetic peptides that correspond to immunogenic epitopes of tumor antigens. The pulsed dendritic cells will then be aliquoted and frozen before shipping back to the site. Patients will have the autologous DCs reinfused intradermally. A control group will receive unpulsed autologous DC. Patients will be randomized by age in a 2:1 ratio to ICT-107 or control.Patients will receive at least four intradermal injections of the ICT-107 vaccine and additional vaccine during a maintenance phase. The primary objective is to compare overall survival (OS) and progression free survival (PFS) in patients when treated with ICT-107 versus Control.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed, initial diagnosis of GBM. Patients must be newly diagnosed with GBM and not yet received chemoradiation.
2. ≥ 18 years of age
3. HLA-A1 or HLA-A2 positive
4. KPS score of ≥ 70%
5. Baseline hematologic studies and chemistry profiles must meet the following criteria:

   Hemoglobin (Hgb) > 9.9 g/dL total granulocyte count > than 1000/mm3 platelet count > 100,000/mm3 blood urea nitrogen (BUN) < 30 mg/dL creatinine < 2 mg/dL alkaline phosphatase (ALP), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 4x upper limit of normal (ULN) prothrombin time (PT) and activated partial thromboplastin time (PTT) ≤ 1.6x control unless therapeutically warranted
6. Female patients of child-bearing potential must have negative serum pregnancy test
7. If not surgically sterile, male and female patients of childbearing age must use double barrier contraception (hormonal; intrauterine device; barrier)
8. Sufficient paraffin embedded tumor sample for analysis MGMT methylation status
9. Written informed consent, Release of Medical Records Form and Health Insurance Portability and Accountability Act (HIPAA) reviewed and signed by patient or legally authorized representatives

Exclusion Criteria:

1. Recurrent disease
2. Radiosurgery including Gamma Knife, linear accelerator based radiosurgery, CyberKnife and placement of Gliadel wafer
3. Presence of any other active malignancy or prior history of malignancy (except for basal cell carcinoma of the skin)
4. Severe pulmonary, cardiac or other systemic disease
5. Congestive heart failure Class III or IV according to New York Heart Association (NYHA)
6. Presence of an acute infection requiring active treatment with antibiotics/antivirals; prophylactic administration is allowed
7. Known history of an autoimmune disorder
8. Known human immunodeficiency virus (HIV) positivity or acquired immunodeficiency syndrome (AIDS) related illness or other serious medical illness
9. Breastfeeding
10. Received any other therapeutic investigational agent within 30 days of enrollment
11. Reduction of steroids (dexamethasone) to a maximum of 2 mg twice a day (BID) prior to the first administration of study vaccine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Gringeri, Ph.D., Study Director — Precision Life Sciences Group
Locations (25):
- United States (25):
  - University of Alabama at Birbingham School of Medicine, South Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Jewish Hospital Medical Center, Louisville, Kentucky
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetss General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - New Jersey Neuroscience Institute, Edison, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Long Island Brain Tumor Center at Neurological Surgery, PC, Great Neck, New York
  - NYU Clinical Cancer Center, New York, New York
  - Weil Cornell Medical College, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Rose Ella Burkhardt Brain Tumor and Neuro Oncology Center, Cleveland, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sammons Cancer Center (Baylor), Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Autologous dendritic cells that have not been pulsed with antigens
  Placebo DC: Autologous dendritic cells (DC) that have not been pulsed with antigens
Period: Overall Study
Arm/Group | ICT-107 | Placebo
Started | 81 | 43
Completed | 75 (Survival is still being assessed) | 42
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ICT-107 | Placebo | Total
Number analyzed (Participants) | 81 | 43 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 29 | 88
  >=65 years | 22 | 14 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 12 | 49
  Male | 44 | 31 | 75
Region of Enrollment [Number; unit: participants]
  United States | 81 | 43 | 124

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The objective is to compare overall survival (OS) in patients when treated with ICT 107 versus Control. OS defined as the time from randomization until date of death or the last date patient known alive (if death is not observed) All randomized patients are included in Intent to Treat analysis
Time Frame: 2 -3 years
Population: Intent to treat include all randomized patients
Measure: Median (95% Confidence Interval); unit: months of survival
Groups:
- ICT-107: Treatment with autologous dendritic cells pulsed with immunogenic peptides
- Control Dendritic Cells: Treatment with autologous dendritic cells not pulsed with immunogenic peptides
Arm/Group | ICT-107 | Control Dendritic Cells
Number analyzed (Participants) | 81 | 43
months of survival | 18.3 [14.9 to 21.2] | 16.7 [12.3 to 23.0]

2. Secondary Outcome: PFS
Description: Secondary Endpoints
  * PFS is defined as the time from randomization until the date of documented progressive disease (PD) or death, whichever occurs first, or last date known alive and progression free if progression or death is not observed.
  * Population is all randomized patients ITT.
Time Frame: 2-3 years
Population: Intent to treat includes all randomized patients
Measure: Median (95% Confidence Interval); unit: months of progression free survival
Arm/Group | ICT-107 | Placebo
Number analyzed (Participants) | 81 | 43
months of progression free survival | 11.2 [8.2 to 13.0] | 9.0 [5.5 to 10.3]
Statistical Analysis 1: Comparison: ICT-107 vs Placebo; Stratified log rank p value stratified for age and MGMT methylation status; Test type: Superiority or Other; p = 0.010, Log Rank — Stratified for age and MGMT methylation status

3. Primary Outcome: Overall Survival in HLA-A2 Patients
Description: Overall survival in a predefined subpopulation. All randomized patients are included in intent to treat analysis.
Time Frame: 2-3 years
Population: Patients with HLA-A2 haplotype
Measure: Median (95% Confidence Interval); unit: months of survival
Arm/Group | ICT-107 | Control
Number analyzed (Participants) | 48 | 29
months of survival | 18.3 [13.2 to 21.1] | 12.9 [10.2 to 19.1]

4. Secondary Outcome: Progression Free Survival in HLA- A2 Patients
Description: Progression Free Survival in a prespecified subpopulation of patients with HLA-A2 haplotype.
  Intent to treat population includes all randomized patients. PFS is defined as the time from randomization until the date of documented progressive disease (PD) or death, whichever occurs first, or last date known alive and progression free if progression or death is not observed
Time Frame: 2-3 yers
Population: HLA-A2 patients
Measure: Median (95% Confidence Interval); unit: months of progression free survival
Arm/Group | ICT-107 | Placebo
Number analyzed (Participants) | 48 | 29
months of progression free survival | 11.2 [6.5 to 14.0] | 7.2 [4.6 to 10.2]
Statistical Analysis 1: Comparison: ICT-107 vs Placebo; Test type: Superiority or Other; p = 0.033, Log Rank — Analyses were stratified for age and MGMT methylation status

ADVERSE EVENTS:
Time Frame: 3 years
Description: Safety population was defined as those receiving at least one dose. This included 80 patients for ICT-107 and 43 patients in the Control group.
Arm/Group | ICT-107 | Placebo
Serious Adverse Events (participants affected / at risk) | 8/80 | 7/43
Other Adverse Events (participants affected / at risk) | 59/80 | 40/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ICT-107 (N=80) | Placebo (N=43)
seizure (Nervous system disorders) | 8 | 7
cerebral edema (Nervous system disorders) | 2 | 1
infection (Infections and infestations) | 4 | 4
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
intracranial hemorrhage (Nervous system disorders) | 4 | 0
increased intracranial pressure (Nervous system disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ICT-107 (N=80) | Placebo (N=43)
convulsion (Nervous system disorders) | 11 | 7
fatigue (General disorders) | 12 | 11
nausea (Gastrointestinal disorders) | 6 | 4
thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3
urinary tract infection (Infections and infestations) | 5 | 2
insomnia (Psychiatric disorders) | 3 | 4
decreased appetite (Metabolism and nutrition disorders) | 2 | 3
upper respiratory tract infection (Infections and infestations) | 0 | 3
white blood cell count decreased (Investigations) | 4 | 0
musular weakness (Musculoskeletal and connective tissue disorders) | 2 | 6
headache (Nervous system disorders) | 2 | 7
hemiparesis (Nervous system disorders) | 4 | 2
partial seizure (Nervous system disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less